CLINICAL TRIAL: NCT02947464
Title: Rapid Maxillary Expansion for Residual Pediatric Obstructive Sleep Apnea After Adenotonsillectomy: a Randomized Controlled Trial
Brief Title: Rapid Maxillary Expansion for Residual Pediatric
Acronym: ERMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, MBarriales, Registered Doctor, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERMES
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard clinical practice
  Interventions: Procedure: Standard clinical practice
- Intervention (Experimental): Standard clinical practice + Rapid Maxillary Expansion
  Interventions: Device: Standard clinical practice + Rapid Maxillary Expansion

INTERVENTIONS:
Procedure: Standard clinical practice — Control weight will be started in obese children to decrease upper airway resistance and airway collapsibility. Close follow-up in order to detect comorbidities.
  Arms: Control
Device: Standard clinical practice + Rapid Maxillary Expansion — Mid-palatal suture osteogenic distraction delivered through a self-activated acrylic intraoral device custom-fit into the children´s palate and maxillary posterior teeth providing a transverse expansion of the dentofacial skeleton.
  Arms: Intervention

SUMMARY:
Randomized Controlled Trial comparing Rapid Maxillary Expansion with Standard Clinical Practice in patients with residual pediatric Obstructive Sleep Apnea Syndrome after adenotonsillectomy.

DETAILED DESCRIPTION:
Cure rate of pediatric Obstructive Sleep Apnea Syndrome (OSAS) after gold-standard-treatment adenotonsillectomy is 50-80%. Treatment alternatives are scarce, poorly effective and based upon low scientific evidence. This means one out of five patients will remain exposed to the well-known neurocognitive, behavioral and quality of life adverse effects of disease.

Rapid Maxillary Expansion, an orthopaedic-orthodontic treatment of pediatric malocclusion, has recently shown promising results in the treatment of pediatric OSAS based upon its effect on craniofacial and upper airway growth, usually limited in these patients.

The investigators propose a randomized, prospective, controlled trial in patients with Pediatric OSAS non-responding to adenotonsillectomy. The aim of the study is to enhance the treatment success rate avoiding morbimortality associated to disease persistence during childhood and development during adult life.

ELIGIBILITY:
Inclusion Criteria:

* Children (boys and girls) between 4 and 9 years of age.
* Residual OSAS after adenotonsillectomy (described as an Apnea Hypopnea Index over 3 objectively measured by means of polysomnography).
* Rapid maxillary expansion indication.
* Parents or tutors sign Informed Consent.

Exclusion Criteria:

* Craniofacial syndromes or neurologic disease diagnosis.
* Adenoid residual hypertrophy occluding >50% nasal airway as measured by means of nasal flexible fiberoptic endoscopy and or tonsillar residual hypertrophy >2 as measured by direct intraoral physical exam.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | During sleep, an average of 10 hours
  Apnea Hypopnea Index (AHI) objectively measured by means of polysomnography.

SECONDARY OUTCOMES:
Sleep-related quality of life | 2 years
  Quality of life as described by OSA-18 questionnaire.
Craniofacial growth | 2 years
  Craniofacial growth by lateral cephalometric radiograph.
Dental arch growth | 2 years
  Dental arch growth as described by Moorrees et al 1969.
Adenotonsillar hypertrophy | 2 years
  Adenotonsillar hypertrophy by nasal flexible fiberoptic endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Fernández-Barriales, Principal Investigator — Basque Health Service
Locations (1):
- Marcos Fernandez-Barriales, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available on reasonable request after completion of the trial